CLINICAL TRIAL: NCT02299427
Title: A Website to Teach Children Safety With Dogs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Schwebel, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD075960 (NIH)
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Child Dog Bite Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dog safety (Experimental): 2 weeks of regular use of website on child dog safety developed for this research
  Interventions: Behavioral: dog safety
- transportation safety (Active Comparator): 2 weeks of regular use of publicly-available website on child transportation safety
  Interventions: Behavioral: transportation safety

INTERVENTIONS:
Behavioral: dog safety — use of dog safety website at home for about 2 weeks
  Arms: dog safety
Behavioral: transportation safety — use of transportation safety website at home for about 2 weeks
  Arms: transportation safety

SUMMARY:
Dog bites result in over 800,000 doctor/ER visits, 6000 hospitalizations, and a dozen deaths each year in the United States. By a large margin, children suffer the highest risk - and children typically are bitten by familiar dogs in familiar places. Several programs exist to reduce pediatric dog bite risk, but few are empirically-supported or theoretically-motivated. None are widely disseminated. This study builds from existing child dog bite prevention programs to develop and then evaluate a website to teach children safe interactions with dogs. The website will be interactive, entertaining, and engaging, allowing children (target ages 4-6) to learn in a technologically-sophisticated and interactive environment. It will be developed based in behavioral theory. Hearkening child development theory, it will teach and permit practice of cognitive skills that develop in early childhood and are critical to safety with dogs: impulse control, perspective taking, and attention to details. Hearkening health behavior change theory, the website will help children and their parents perceive personal vulnerability to bites, recognize normative behavior to protect themselves, and have personal motivation to change previous habits. Overarching the website design will be goals to create an engaging and entertaining environment, and to facilitate cognitive and behavioral change on the part of both child and parent via multiple mechanisms. Besides teaching children, the website will educate parents via an innovative messaging system triggered by child attainment of points and "skill levels".

Following website development, an evaluation study will investigate usability and efficacy of the website using a repeated measures pre-test, post-test experimental design. 68 children ages 4-6 will be recruited, complete a pre-intervention assessment evaluating knowledge and behavior relevant to dog safety via multiple methods, and then be randomly assigned to use either the newly-developed dog safety website or a control pedestrian safety website at home over the subsequent 2 weeks. Frequent reminders will encourage website use. Following the 2-week period, all children will return for a post-intervention assessment battery to evaluate knowledge and behavior change. Data will be analyzed using descriptive and inferential statistics, with primary hypotheses tested using linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* parent and child speak English,
* exposure to dogs with some frequency,
* internet access at home

Exclusion Criteria:

* physical or disability preventing valid participation in study

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
After primary analyses will completed, will provide de-identified data to qualified users who contact us.

REFERENCES:
- [Background] Schwebel DC, McClure LA, Severson J. Evaluating a website to teach children safety with dogs. Inj Prev. 2015 Feb;21(1):e2. doi: 10.1136/injuryprev-2014-041286. Epub 2014 May 28. PMID 24871960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dog Safety | Transportation Safety
Started | 35 | 34
Completed | 12 | 31
Not Completed | 23 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — not adherent to dog website use | 21 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dog Safety | Transportation Safety | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.0 (0.6) | 5.1 (0.6) | 5.1 (.6)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 22 | 36
  Male | 21 | 12 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 6 | 10 | 16
  Caucasian | 27 | 19 | 46
  Other | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Children's Behavior With Dogs on Standardized Objective Scale
Description: Coded behavior using objective criteria during a semi-structured interaction with a live therapy dog. Specifically, we examined behavioral patterns for 15 tasks/activities/decisions the child made with the live dog. Sample tasks were when and how the child touched the dog, the extent to which the child was close or intimate to the dog, whether the child handled the dog's toys, and whether the child interrupted the dog during its "rest time". 7 of those hung together in factor analysis. Those 7 were standardized and then averaged to create the scale. It was transformed with linear transformation so all values are positive. Higher numbers indicate higher risk-taking. Theoretically the scale is 0-infinity; in practice most children scored between 0-4. The individual items had an average intercorrelation of .50 and Cronbach's alpha of .65.
Time Frame: post-intervention (about 2 weeks after pre-intervention assessment)
Population: In the dog safety group, only children with known noncompliance were analyzed for this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dog Safety | Transportation Safety
Number analyzed (Participants) | 12 | 34
units on a scale | 1.4 (.5) | 1.6 (.8)

2. Primary Outcome: Simulated Behavior With Dogs on Standardized Objective Scale
Description: Coded behavior in dollhouse simulation. Specifically, in 7 simulated scenarios using a dollhouse that included child and dog characters, furniture, yard, etc., children heard a scene and explained/used the dolls to act what would happen next. For example, the experimenter acted a child doll playing in the kitchen near dog food and the doll dog entered, saw the child, and approached the food bowl. The experimenter said, "[Child's Name] is playing around in the kitchen near [Dog name's] food. [Dog's name] comes into the kitchen and sees [Child's Name] near his/her food bowl making him/her upset and start to growl. What will happen next?" The task was coded using objective coding criteria to score the child's response as safe (1 point), safe but not optimal (0.5 points), or unsafe (0 points). Scores across the 7 scenarios were summed to yield a single score; possible range = 0=7. Higher scores indicate better safety. Inter-rater reliability on 30% of the sample was good; kappa = .90.
Time Frame: post-intervention (about 2 weeks after pre-intervention assessment)
Population: In the dog safety group, only children with known noncompliance were analyzed for this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dog Safety | Transportation Safety
Number analyzed (Participants) | 12 | 34
units on a scale | 3.0 (2.0) | 3.6 (2.1)

ADVERSE EVENTS:
Groups:
- Dog Safety: 2 weeks of regular use of website on child dog safety developed for this research
  dog safety: use of dog safety website at home for about 2 weeks
  There is a discrepancy in participants at risk compared to the participant flow module because some children were not compliant to the intervention. They did not use the internet website and therefore were excluded from analyses. They did not have adverse events; they merely were not exposed to the intervention and therefore were excluded from analysis.
Arm/Group | Dog Safety | Transportation Safety
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dog Safety (N=35) | Transportation Safety (N=34)
adverse medical or social situations (Social circumstances) | 0 (0) | 0 (0) — no adverse events occurred; we monitored increased risk for injury, negative medical consequences including dog bites, breach of confidentiality, and other adverse situations to participants and their families

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No